CLINICAL TRIAL: NCT04444336
Title: Information Sources and Their Relationship to Depressive and Anxiety Symptoms During the COVID-19 Pandemic: A Network Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Oslo (Other)
Collaborators: Modum Bad (Other)
Responsible Party: Principal Investigator, Omid V. Ebrahimi, Principal investigator, University of Oslo
Other Study IDs: REK125510-16
Record Dates: First submitted 2020-06-21; First posted 2020-06-23 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Cross-sectional study examining the impact of information sources to obtain information about COVID-19 on depression and anxiety symptoms — Cross-sectional study examining the impact of information sources to obtain information about COVID-19 on depression and anxiety symptoms

SUMMARY:
This study aims to investigate the association between the use different information sources to obtain information about the COVID-19 pandemic and symptoms of psychopathology (i.e., depression and anxiety).

Research Question:

How central are different sources of information used to obtain knowledge about the COVID-19 pandemic in network along with depressive and anxiety symptoms? Which sources of information are most strongly connected to different symptoms of depression and anxiety? Staying away from information will be measured in the present study. As avoidance is a type of safety behavior in anxiety disorders, we are further eager to investigate the centrality of this behavior in the network. Furthermore, multiple studies using latent-variable paradigms have established a relationship between sum-scores of depression and social anxiety use in general. We are further interested in examining this potential link more thoroughly and detailed in the present network study. The findings of this study, although they will be cross-sectional and require further examination in studies with temporal data structure, will be an important and interesting starting point giving initial ideas about potential mechanisms that may be involved in use of information sources in pandemics and mental health

DETAILED DESCRIPTION:
Research Question 1:

How central are different sources of information used to obtain knowledge about the COVID-19 pandemic in network along with depressive and anxiety symptoms? Which sources of information are most strongly connected to different symptoms of depression and anxiety?

Staying away from information will be measured in the present study. As avoidance is a type of safety behavior in anxiety disorders, the investigators are further eager to investigate the centrality of this behavior in the network. Furthermore, multiple studies using latent-variable paradigms have established a relationship between sum-scores of depression and social anxiety use in general. The investigators are further interested in examining this potential link more thoroughly and detailed in the present network study. The findings of this study, although they will be cross-sectional and require further examination in studies with temporal data structure, will be an important and interesting starting point giving initial ideas about potential mechanisms that may be involved in use of information sources in pandemics and mental health.

Statistical analysis:

The estimated network will consist of 23 items (9: PHQ-9; 7: GAD-7; 7: information sources to obtain information about COVID-19). The network will be estimated using the R package qgraph (Epskamp et al., 2012). Network stability and accuracy tests will be conducted using R package bootnet (Epskamp, et al., 2018). An undirected partial correlation network will be estimated, resulting in associations between each pair of symptoms controlling for all other associations among symptoms. Centrality indices will be reported. The appropriate correlation method will be applied following an assessment of the data (e.g., with regards to possible skewness).

The network will further be regularized using Graphical Least Absolute Shrinkage and Selection Operator (GLASSO), with Extended Bayes Information Criterion (EBIC). The tuning parameter will be set to 0.5, as is recommended practice. Centrality table and plots will be depicted, and difference test of edges conducted.

Additionally, the investigators will investigate differences in network structure across major demographic subgroups in the sample (e.g., gender). All analyses and questions addressed in the forthcoming paper that are not pre-specified in this pre-registered protocol will be defined as exploratory.

The sources of information include: 1) National television and radio channels; 2) national and regional, and local newspapers; 3) Use of social media for information; 4) use of blogs, podcasts, forums or other Internet sources; 5) information obtained from peers (i.e., friends and family); 6) Other sources of information; 7) actively staying away from information.

Inference criteria:

p < 0.05 to determine significance.

Sample size and power calculation:

Following power analysis guidelines by Fried & Cramer (2017), it is recommended that the number of participants are three times larger than the number of estimated parameters. However, more conservative recommendations by Roscoe (1975) for multivariate research, recommends sample size that is ten times larger than the number of estimated parameters. The network to be constructed for this study consists of 7 anxiety items (GAD-7), 9 depression symptom items (PHQ-9), and the 7 pre-specified items above concerning medium of information and extent of use. Consequently, the network consists of 23 items. 23x(23-1)/2 x 3 = at least 759 participants (according to guidelines by Fried & Cramer, 2017). Thus, following these two approaches respectively, between 759 to 2530 participants are required. Data will be collected for three weeks, and participants are based on a representative sample of Norwegian adults with equal opportunity to partake in the study following providing digital consent.

Missing data:

The TSD system (Services for Sensitive Data), a platform used in Norway to store person-sensitive data verifies participants officially through a kind of national ID number to give them full right to withdraw their data at any time, following the European GDPR (General Data Protection Regulation) laws. Accordingly, participants are allowed to withdraw their own data at any time. The survey includes mandatory fields of response. Participation is voluntarily, and withdrawal of any provided data is possible at any moment. The investigators do not expect participants to withdraw their data and thus expect no missing data. However, if participants do withdraw their data, the investigators will conduct state-of-art missing data analysis and investigate whether data is missing at random.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants are all adults including those of 18 years and above,
* Who are currently living in Norway and thus experiencing identical NPIs, and
* Who will provide digital consent to partake in the study.

Exclusion Criteria:

* Children and adolescents (individuals below 18)
* Adults not residing in Norway during the measurement period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Both Biological Sex and self-representation of gender are measured
Study Population: All adults above 18 years residing in Norway and thus experiencing identical mitigation protocols are invited to participate the study, reached through a random digital sample, providing consent digitally.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-06-22 (Estimated); Primary Completion 2020-07-13 (Estimated); Study Completion 2020-07-13 (Estimated)

PRIMARY OUTCOMES:
The Patient Health Questionnaire 9 | Data is set to be collected starting from 22nd of June until enough data has been collected. The data collection period will last no longer than three weeks.
  The Patient Health Questionnaire 9 (PHQ-9; Kroenke, Spitzer & Williams, 2001) is used to measure symptoms of depression in accordance with the diagnostic criteria for major depressive disorder. The questionnaire consists of nine items where each is scored on a four-point Likert scale (0-3), with the range of scores from 0 to 27. Higher scores indicate greater depression severity, and scores above 10 are considered as the cut-off that indicating that the patient is within the depressive area.
Generalized Anxiety Disorder 7 | Data is set to be collected starting from 22nd of June until enough data has been collected. The data collection period will last no longer than three weeks.
  The Generalized Anxiety Disorder 7 (GAD-7; Spitzer, Kroenke, Williams & Löwe, 2006) is a questionnaire consisting of seven items measuring symptoms of anxiety and worry. The items are scored on a four-point Likert scale (0-3), with the scores ranging from 0 to 21. Specific cut-off for Norwegian samples have been found yielding a cut-off of 8 and above for high sensitivity and specificity (Johnson, Ulvenes, Øktedalen & Hoffart, 2019).

CONTACTS AND LOCATIONS:
Overall Officials: Omid Ebrahimi, Double PhD Candidate, Principal Investigator — University of Oslo; Asle Hoffart, PhD, Principal Investigator — Modum Bad; Sverre Urnes Johnson, PhD, Principal Investigator — University of Oslo

REFERENCES:
- [Background] Fried EI, Cramer AOJ. Moving Forward: Challenges and Directions for Psychopathological Network Theory and Methodology. Perspect Psychol Sci. 2017 Nov;12(6):999-1020. doi: 10.1177/1745691617705892. Epub 2017 Sep 5. PMID 28873325
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171